CLINICAL TRIAL: NCT02283645
Title: Efficacy and Safety of 3% Minoxidil Lotion for Chest Hair Enhancement : A Randomized, Double-blind, Placebo-controlled Study
Brief Title: Efficacy and Safety of 3% Minoxidil Lotion for Chest Hair Enhancement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mae Fah Luang University Hospital (Other)
Responsible Party: Principal Investigator, Chuchai TANGLERTSAMPAN, MD, Assitant Professor, Mae Fah Luang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REH-57080
Record Dates: First submitted 2014-11-02; First posted 2014-11-05 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Chest Hair Enhancement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minoxidil (Experimental): 3% Minoxidil lotion is applied twice daily to the chest.
  Interventions: Drug: 3 % minoxidil lotion
- Placebo (Placebo Comparator): Placebo lotion is applied twice daily to the chest.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 3 % minoxidil lotion
  Arms: Minoxidil
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine efficacy and safety of 3% minoxidil lotion for chest hair enhancement.

ELIGIBILITY:
Inclusion Criteria:

* healthy male

Exclusion Criteria:

* serious underlying diseases
* history of chest/ hair treatment before 6 months
* history of surgery or trauma on chest area.
* history of minoxidil allergy

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
The change of global photographic assessment after 20 weeks from baseline | baseline and 20 weeks

SECONDARY OUTCOMES:
The change in number of hairs after 20 weeks from baseline | baseline and 20 weeks

OTHER OUTCOMES:
The change of hair diameter after 20 weeks from baseline | baseline and 20 weeks
Number of participants with adverse events | baseline and 20 weeks
Patient satisfaction by self-assessment questionnaires | baseline and 20 weeks

REFERENCES:
- [Result] Lee S, Tanglertsampan C, Tanchotikul M, Worapunpong N. Minoxidil 2% lotion for eyebrow enhancement: a randomized, double-blind, placebo-controlled, spilt-face comparative study. J Dermatol. 2014 Feb;41(2):149-52. doi: 10.1111/1346-8138.12275. Epub 2013 Nov 8. PMID 24471459
- [Result] Suwanchatchai W, Tanglertsampan C, Pengsalae N, Makornwattana M. Efficacy and safety of bimatoprost 0.03% versus minoxidil 3% in enhancement of eyebrows: a randomized, double-blind, split-face comparative study. J Dermatol. 2012 Oct;39(10):865-6. doi: 10.1111/j.1346-8138.2012.01579.x. Epub 2012 May 17. No abstract available. PMID 22594928
- [Result] Tanglertsampan C. Efficacy and safety of 3% minoxidil versus combined 3% minoxidil / 0.1% finasteride in male pattern hair loss: a randomized, double-blind, comparative study. J Med Assoc Thai. 2012 Oct;95(10):1312-6. PMID 23193746